CLINICAL TRIAL: NCT02587234
Title: Driving Neuroplasticity With Nerve Stimulation and Modified Constraint-Induced Therapy
Brief Title: Driving Neuroplasticity With Nerve Stimulation and Modified CIT
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of Kentucky (Other)
Responsible Party: Principal Investigator, Lumy Sawaki, Associate Professor, University of Kentucky
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: R03HD049408 (NIH)
Record Dates: First submitted 2015-10-23; First posted 2015-10-27 (Estimated); Results first posted 2017-07-14 (Actual); Last update posted 2023-09-13 (Actual); Status verified 2023-09

CONDITIONS: Stroke; Cerebrovascular Accident
Keywords: motor recovery; chronic; human; sensory; afferent input; motor training
MeSH Terms: conditions — Stroke; Bronchiolitis Obliterans Syndrome

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Active (Experimental): 2 hours of active peripheral nerve stimulation paired with 4 hours of intensive task-oriented upper extremity training
  Interventions: Device: peripheral nerve stimulation
- Sham PNS (Sham Comparator): 2 hours of sham peripheral nerve stimulation paired with 4 hours of intensive task-oriented upper extremity training
  Interventions: Device: peripheral nerve stimulation

INTERVENTIONS:
Device: peripheral nerve stimulation — Non-invasive stimulation of median, ulnar and radial nerves

SUMMARY:
The investigators proposed to evaluate the effectiveness of sustained peripheral nerve stimulation (PNS) to enhance the therapeutic effects of a modified form CIT (mCIT).

DETAILED DESCRIPTION:
Stroke is one the most devastating and prevalent diseases, but efforts to limit the amount of tissue damaged in the acute phase have been disappointing, highlighting the need for effective therapeutic interventions after neurologic damage has occurred. A major goal of the research in stroke rehabilitation is to harness the capacity of the brain to reorganize after neurologic damage has occurred and thus ultimately lead to successful recovery of function. Data from animal and human models have suggested that sensory input plays an important role in motor output, possibly by influencing cortical plasticity. However, in spite of the advances to date, little is known about the extent to which sensory input in the form of peripheral nerve stimulation can be successfully combined to physical training. A new emerging approach called constraint-induced therapy (CIT) is an intensive functional motor training and has produced promising results in the field of stroke rehabilitation. CIT involves restraining the unaffected arm with a sling or glove combined with intense task-oriented therapy of the affected side for six hours daily during 2 weeks. This pilot study will evaluate the effectiveness of sustained peripheral nerve stimulation coupled with functional motor training to improve hand motor function. While the functional motor training follows identical principles of CIT, the length of daily training will be shortened to 4 hours daily and thus the investigators will refer in this proposal as a modified CIT. Preliminary data for this study demonstrated that peripheral nerve stimulation results in increased cortical motor excitability in normal subjects. In addition, learning and use-dependent plasticity can be substantially enhanced by a single session of 2 hours of peripheral nerve stimulation in chronic stroke patients. The goal of this study is to test the hypothesis that stroke patients treated with upper extremity peripheral nerve stimulation preceding CIT (intervention group) will have improved hand motor function compared to a group receiving lower extremity peripheral nerve stimulation and CIT (control group).

ELIGIBILITY:
Inclusion Criteria:

* Chronic stroke patients
* Single stroke
* Chronic (more than 12 months after from stroke)
* At least 21 years old, but there is no upper age range for this project.
* Participants must be able to extend the affected metacarpophalangeal joints at least 10° and the wrist 20°.

Exclusion Criteria:

* History of carpal tunnel syndrome and conditions that commonly cause peripheral neuropathy, including diabetes, uremia, or associated nutritional deficiencies
* History of head injury with loss of consciousness, severe alcohol or drug abuse, psychiatric illness
* Within 3 months of recruitment, use of drugs known to exert detrimental effects on motor recovery
* Cognitive deficit severe enough to preclude informed consent
* Positive pregnancy test or being of childbearing age and not using appropriate contraception
* Participants with history of untreated depression.

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2006-11; Primary Completion 2010-02 (Actual); Study Completion 2012-04 (Actual)

REFERENCES:
- [Derived] Carrico C, Chelette KC 2nd, Westgate PM, Salmon-Powell E, Nichols L, Sawaki L. Randomized Trial of Peripheral Nerve Stimulation to Enhance Modified Constraint-Induced Therapy After Stroke. Am J Phys Med Rehabil. 2016 Jun;95(6):397-406. doi: 10.1097/PHM.0000000000000476. PMID 26945226

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Active | Sham PNS
Started | 11 | 10
Completed | 10 | 7
Not Completed | 1 | 3
Not completed — Withdrawal by Subject | 1 | 1
Not completed — Lost to Follow-up | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- Active PNS: 2 hours of active peripheral nerve stimulation paired with 4 hours of intensive task-oriented upper extremity training
  peripheral nerve stimulation: Non-invasive stimulation of median, ulnar and radial nerves
- Total: Total of all reporting groups
Arm/Group | Active PNS | Sham PNS | Total
Number analyzed (Participants) | 11 | 10 | 21
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: Age calculations exclude the subject from the Active PNS group who withdrew during the interventions and the subject from the Sham PNS group who withdrew during the interventions.
  years
    number analyzed (Participants) | 10 | 9 | 19
    (all) | 56.7 (8.6) | 54.6 (10.2) | 55.7 (9.2)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: Numbers do not include the 2 subjects who withdrew prior to completing the interventions.
  Participants
    number analyzed (Participants) | 10 | 9 | 19
    Female | 7 | 3 | 10
    Male | 3 | 6 | 9

OUTCOME MEASURES:

1. Primary Outcome: Change in Wolf Motor Function Test (WMFT), Timed Portion
Description: Score at post-intervention minus score at baseline, score at 1-month follow-up minus score at baseline
Time Frame: baseline, post-intervention, 1-month follow-up
Population: Two subjects in the Sham PNS group were lost to follow-up.
Measure: Mean (95% Confidence Interval); unit: log(seconds)
Arm/Group | Active PNS | Sham PNS
Number analyzed (Participants) | 10 | 9
log(seconds)
  Post-intervention minus baseline | -0.36 [-0.45 to -0.27] | -0.18 [-0.28 to -0.07]
  1-month follow-up minus baseline: number analyzed (Participants) | 10 | 7
  1-month follow-up minus baseline | -0.37 [-0.51 to -0.22] | -0.15 [-0.29 to -0.01]

2. Secondary Outcome: Change in Fugl Meyer Assessment Motor Score
Description: Score at post-intervention minus score at baseline, score at 1-month follow-up minus score at baseline. The scores can range from 0 to 66, with higher scores indicating better performance. The scores are calculated by summing the scores to the 33 individual tasks.
Time Frame: baseline, post-intervention, 1-month follow-up
Population: Two subjects from the Sham PNS group were lost to follow-up.
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Active PNS | Sham PNS
Number analyzed (Participants) | 10 | 9
units on a scale
  Post-intervention minus baseline | 10.2 [7.44 to 12.96] | 5.6 [2.34 to 8.77]
  1-month follow-up minus baseline: number analyzed (Participants) | 10 | 7
  1-month follow-up minus baseline | 12.5 [7.52 to 17.48] | 6.3 [2.96 to 9.61]

3. Secondary Outcome: Change in Action Research Arm Test (ARAT)
Description: Values given are score at post-intervention minus score at baseline, score at 1-month follow-up minus score at baseline.
  The ARAT's is a 19 item measure divided into 4 sub-tests (grasp, grip, pinch, and gross arm movement).
  Performance on each item is rated on a 4-point ordinal scale ranging from:
  3: Performs test normally 2: Completes test, but takes abnormally long or has great difficulty
  1: Performs test partially 0: Can perform no part of test The maximum score on the ARTS is 57 points (possible range 0 to 57).
Time Frame: baseline, post-intervention, 1-month follow-up
Population: Two subjects from the Sham PNS group were lost to follow-up.
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Active PNS | Sham PNS
Number analyzed (Participants) | 10 | 9
units on a scale
  Post-intervention minus baseline | 9.6 [5.64 to 13.57] | 3.67 [2.28 to 5.05]
  1-month follow-up minus baseline | 11.1 [5.43 to 16.77] | 4.43 [2.67 to 6.19]

ADVERSE EVENTS:
Arm/Group | Active PNS | Sham PNS
Serious Adverse Events (participants affected / at risk) | 0/11 | 0/10
Other Adverse Events (participants affected / at risk) | 1/11 | 0/10
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Active PNS (N=11) | Sham PNS (N=10)
Fall (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) — Subject sustained a fall at home during the intervention period of the study. The subject was evaluated by a doctor not associated with the study and no fractures or major trauma was detected. The event was determined to not be related to the study.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No